CLINICAL TRIAL: NCT03916952
Title: The Effects of Guarding on the Outcomes of the Six Minute Walk Test
Status: Completed | Type: Observational
Sponsor: Concordia University, St. Paul (Other)
Responsible Party: Principal Investigator, Kristin Lefebvre, Principle investigator, Concordia University, St. Paul
Other Study IDs: ConcordiaUStPau
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Functional Capacity; Physical Activity; Rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Walk Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy younger: All participants between 18 and 65 years of age that completed the test
  Interventions: Diagnostic Test: Six Minute Walk Test
- Healthy older: All participants > 65 years of age that completed the test
  Interventions: Diagnostic Test: Six Minute Walk Test

INTERVENTIONS:
Diagnostic Test: Six Minute Walk Test — The patients walked as far as possible for 6 minutes--over two separate trials. In one trial, an examiner walked with the participant. In the second trial, the participant walked independently. A paired T test was performed to see if there was a significant difference in the distance walked or gait speed between the trials.

SUMMARY:
This study was designed to determine if walking with a healthy individual during the 6 minute walk test significantly influenced the outcome of the test.

DETAILED DESCRIPTION:
Introduction: The American Thoracic Society recommends not walking with the patient or client during the Six Minute Walk Test (6MWT). However, this recommendation raises safety concerns for individuals at increased risk of falls. Given the recommendations and concerns, the effects of guarding during the 6MWT has not been investigated. Purpose: The purpose of this study was to determine if guarding during the 6MWT affected gait speed and distance walked. Methods: Participants were randomized into a 'guarded first' vs 'guarded second' condition. Data were analyzed using a one-sample t-test, Pearson Correlation Coefficients, Intraclass Correlation Coefficients (ICC), and Bland Altman plots to assess differences and relationships for gait speed and distance walked between the guarded and unguarded trials.

ELIGIBILITY:
Inclusion Criteria:

Young Group

* Between 18 and 50 years of age
* Independent with ambulation such that no physical assistance was required during the 6MWT
* No pertinent acute or chronic medical conditions.

Older adult group

* 50 years of age or older Ambulatory without requiring physical assistance Intact cognition as determined by achieving a score of 24 on the Mini Mental Status Exam
* Stable balance by scoring a minimum of 18cm (7 inches) on the Functional Reach Test

Exclusion Criteria:

* All Participants:
* Unstable angina
* History of myocardial infarction 30 days prior to the study
* Resting heart rate greater than 120 beats per minute
* Resting systolic blood pressure greater than 180 mmHg
* Resting diastolic blood pressure greater than 100 mmHg
* Symptoms were reported or observed that were consistent with low blood pressure
* Recent injury, surgery or medical procedure.
* Older Participants:
* Functional Reach Test (<18cm or 7 inches)
* Mini Mental Exam (score < 24).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Boxes for Male, Female and Other were provided on demographic form
Study Population: The study population was average age of 24 in the younger group and 71.2 in the older group. The population was 134 female to 69 males. The sample population was primarily Caucasian (89%). Mean BMI of the younger group was 24.1 and the older group 26.4.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2017-06-11 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Distance Walked | 6 Minutes
  How far the patient was able to ambulate
Gait Speed | 6 Minutes
  How fast the patient was able to ambulate

CONTACTS AND LOCATIONS:
Locations (1):
- Widener University, Chester, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casanova C, Celli BR, Barria P, Casas A, Cote C, de Torres JP, Jardim J, Lopez MV, Marin JM, Montes de Oca M, Pinto-Plata V, Aguirre-Jaime A; Six Minute Walk Distance Project (ALAT). The 6-min walk distance in healthy subjects: reference standards from seven countries. Eur Respir J. 2011 Jan;37(1):150-6. doi: 10.1183/09031936.00194909. Epub 2010 Jun 4. PMID 20525717
- [Background] Bohannon RW, Crouch R. Minimal clinically important difference for change in 6-minute walk test distance of adults with pathology: a systematic review. J Eval Clin Pract. 2017 Apr;23(2):377-381. doi: 10.1111/jep.12629. Epub 2016 Sep 4. PMID 27592691
- [Background] Wise RA, Brown CD. Minimal clinically important differences in the six-minute walk test and the incremental shuttle walking test. COPD. 2005 Mar;2(1):125-9. doi: 10.1081/copd-200050527. PMID 17136972
- [Background] Bohannon RW. Comfortable and maximum walking speed of adults aged 20-79 years: reference values and determinants. Age Ageing. 1997 Jan;26(1):15-9. doi: 10.1093/ageing/26.1.15. PMID 9143432
- [Background] Chetta A, Zanini A, Pisi G, Aiello M, Tzani P, Neri M, Olivieri D. Reference values for the 6-min walk test in healthy subjects 20-50 years old. Respir Med. 2006 Sep;100(9):1573-8. doi: 10.1016/j.rmed.2006.01.001. Epub 2006 Feb 7. PMID 16466676
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Bland JM, Altman DG. Agreement between methods of measurement with multiple observations per individual. J Biopharm Stat. 2007;17(4):571-82. doi: 10.1080/10543400701329422. PMID 17613642
- [Background] Cicchetti D, Bronen R, Spencer S, Haut S, Berg A, Oliver P, Tyrer P. Rating scales, scales of measurement, issues of reliability: resolving some critical issues for clinicians and researchers. J Nerv Ment Dis. 2006 Aug;194(8):557-64. doi: 10.1097/01.nmd.0000230392.83607.c5. PMID 16909062
- [Background] Stevens D, Elpern E, Sharma K, Szidon P, Ankin M, Kesten S. Comparison of hallway and treadmill six-minute walk tests. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1540-3. doi: 10.1164/ajrccm.160.5.9808139. PMID 10556117
- [Background] de Almeida FG, Victor EG, Rizzo JA. Hallway versus treadmill 6-minute-walk tests in patients with chronic obstructive pulmonary disease. Respir Care. 2009 Dec;54(12):1712-6. PMID 19961638
- [Background] Bansal V, Hill K, Dolmage TE, Brooks D, Woon LJ, Goldstein RS. Modifying track layout from straight to circular has a modest effect on the 6-min walk distance. Chest. 2008 May;133(5):1155-60. doi: 10.1378/chest.07-2823. Epub 2008 Feb 8. PMID 18263673
- [Background] Smith MD, Chang AT, Seale HE, Walsh JR, Hodges PW. Balance is impaired in people with chronic obstructive pulmonary disease. Gait Posture. 2010 Apr;31(4):456-60. doi: 10.1016/j.gaitpost.2010.01.022. Epub 2010 Mar 4. PMID 20206529
- [Background] Lederer DJ, Arcasoy SM, Wilt JS, D'Ovidio F, Sonett JR, Kawut SM. Six-minute-walk distance predicts waiting list survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2006 Sep 15;174(6):659-64. doi: 10.1164/rccm.200604-520OC. Epub 2006 Jun 15. PMID 16778159
- [Background] VanWagner LB, Uttal S, Lapin B, Lee J, Jichlinski A, Subramanian T, Heldman M, Poole B, Bustamante E, Gunasekaran S, Tapia CS, Veerappan A, Wong SY, Levitsky J. Use of Six-Minute Walk Test to Measure Functional Capacity After Liver Transplantation. Phys Ther. 2016 Sep;96(9):1456-67. doi: 10.2522/ptj.20150376. Epub 2016 Apr 7. PMID 27055540